CLINICAL TRIAL: NCT02800928
Title: Does CERC-501 Attenuate Stress-precipitated Smoking Lapse?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Office of Research on Women's Health (ORWH) (NIH); Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sherry McKee, Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1602017291; P50DA033945 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-06-15 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CERC-501 (Experimental): Administered orally once daily, 10mg daily, 8 days
  Interventions: Drug: CERC-501
- Placebo (Placebo Comparator): Administered orally daily, 8 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CERC-501 — CERC-501
  Arms: CERC-501
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Crossover Design Study of CERC-501 in a Human Laboratory Model of Stress-precipitated Smoking Behavior.

DETAILED DESCRIPTION:
The study will be performed in subjects who are heavy cigarette smokers currently not seeking treatment for tobacco use disorder.

The study is a crossover design study (within-subject analysis), which allows for subjects to be their own control.

Each period of the crossover consists of a 7-day out-patient treatment period followed by a single out-patient testing day on Day 8. Subjects will participate in a laboratory session following the McKee Stress-Smoking Lapse Test. Upon completion, subjects will undergo a 7 day washout period followed by the second period of the crossover design and a 7-day follow-up visit.

ELIGIBILITY:
Inclusion Criteria

1. Provides written informed consent and agrees to complete required clinic visits
2. Male or female 21 to 60 years of age inclusive
3. Body mass index (BMI) 18.5 to 40 kg/m2 inclusive
4. Smokes at least 10 cigarettes per day on average for the past 6 months
5. Fagerstrom score ≥3 at screening
6. Currently not seeking smoking cessation therapy
7. Urine dip test for cotinine concentration >150 ng/mL
8. In otherwise good general health without any unstable medical conditions (as determined by medical history, medication history, physical examination, 10- or 12 lead ECG, vital signs, and clinical laboratory testing)
9. Able to read, write, and speak English
10. Females must be either:

    1. Post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile -or-
    2. Women of childbearing potential (WOCBP) must meet the criteria below:

    i. Uses an acceptable double-barrier method of contraception as determined by the Investigator -and- ii. Is not lactating, has a negative serum beta human chorionic gonadotropin pregnancy test at screening and a negative urine pregnancy test prior to dosing on Days 1 and 8 of each treatment period.
11. Male subjects must agree to use a condom if partner is of childbearing potential

Exclusion Criteria

1. Have used tobacco or other nicotine containing products other than cigarettes (e.g., nicotine patches, pipe, cigars, snuff, chewing tobacco or e-cigarettes) within the past 30 days
2. Any substance use disorder other than nicotine or caffeine as assessed by the Structured Clinical Interview-IV Axis I Disorders (SCID) for Diagnostic and Statistical Manual of Mental Disorders (DSM)
3. Current neurological conditions that interfere with study conduct, assessment or treatment in any significant fashion
4. Any lifetime history of bipolar I, II; schizophrenia or any other psychotic disorders; personality disorders, impulse control disorders as assessed by the SCID-IV
5. Current psychiatric conditions that interfere with study conduct, assessment, or treatment in any significant fashion, such as major depressive disorder (MDD), eating disorders, post-traumatic stress disorder, etc. We will screen for worsening of symptoms of depression and/or suicidality at each medication appointment and lab sessions by having participants complete the Beck Depression Inventory (BDI) and the Columbia-Suicide Severity Rating Scale (C-SSRS). If there is a worsening of symptoms of depression and/or suicidality, the participants will speak a licensed psychologist for evaluation.
6. Recent active or past history of gastric disease such as peptic ulcer disease, gastritis, upper gastrointestinal bleeding, or any gastrointestinal malignancy or precancerous condition
7. Active, comorbid disease that might limit the ability of the subject to participate in the study as determined by the Study MD (i.e., poorly controlled diabetes mellitus, congestive heart failure, etc.)
8. Clinically significant clinical laboratory test taken during screening
9. Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2 times the upper limit of normal (ULN)
10. Human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C positive as determined by serology testing at Screening
11. Positive ethanol breath test at screening or prior to dosing on Days 1 and 8 of each treatment period
12. Positive urine drug test at screening or and/or prior to dosing on Days 1 and 8 of each treatment period except for cannabis
13. History of severe allergies or multiple adverse drug reactions
14. Known hypersensitivity to CERC-501
15. Current use of a proton pump inhibitor or histamine 2 blocker
16. Use of any investigational medication within 2 months prior to the start of this study or scheduled to receive an investigational drug other than the study drug during the course of this study
17. Current use of any psychoactive medications including: antipsychotics, benzodiazepines, mood stabilizers, selective serotonin reuptake inhibitor/serotonin norepinephrine reuptake inhibitor (SSRI/SNRI) or other antidepressants mood stabilizers

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a cross-over design. Medication arms are within-subject.
Groups:
- Treatment First: Administered orally once daily, 10mg daily, 8 days
  CERC-501: CERC-501
  7 day wash-out
  Administered orally once daily, placebo, 8 days
  Order of placebo/CERC-501 counterbalanced
- Placebo First: Administered orally once daily, placebo, 8 days FIRST
  7 day wash-out
  Administered orally once daily, CERC-501: CERC-501 10mg daily, 8 days SECOND
Period: Overall Study
Arm/Group | Treatment First | Placebo First
Started | 9 | 8
Completed | 7 | 6
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Administered orally once daily, 10mg daily, 8 days
  CERC-501: CERC-501
  7 day wash-out
  Administered orally once daily, placebo
  Order of placebo/CERC-501 counterbalanced
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.18 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 16.24 (3.90)

OUTCOME MEASURES:

1. Primary Outcome: Latency
Description: Latency (in minutes and seconds) to time of first cigarette smoking during the delay period
Time Frame: 50 min
Population: 13 subjects completed study (i.e., completed both CERC-501 and Placebo periods in this cross over design).
Measure: Mean (Standard Error); unit: minutes
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 13 | 13
minutes | 24.56 (6.40) | 26.64 (6.62)

2. Primary Outcome: Number of Cigarettes Smoked
Description: Number of cigarettes smoked during the self administration period
Time Frame: 60 min
Measure: Mean (Standard Error); unit: number of cigarettes
Arm/Group | CERC-501 | Placebo
Number analyzed (Participants) | 13 | 13
number of cigarettes | 1.67 (0.28) | 1.92 (0.25)

ADVERSE EVENTS:
Time Frame: 8 days
Description: SAFTEE assessment.
  In total 16 subjects were exposed to CERC-501 and are included in adverse event analysis. In total 15 subjects were exposed to placebo and are included in the adverse event analysis. This is a cross-over design.
Arm/Group | CERC-501 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 3/16 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CERC-501 (N=16) | Placebo (N=15)
headache (General disorders) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
insomnia (General disorders) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT02800928/Prot_SAP_000.pdf